CLINICAL TRIAL: NCT00508859
Title: Maintenance Study for Adolescent Depression
Acronym: MTAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Medical Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0831997
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Depression
Keywords: depression; adolescents; maintenance treatment; antidepressant
MeSH Terms: conditions — Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active, 1 (Experimental): sertraline
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sertraline — maintenance treatment with sertraline
  Other Names: zoloft
  Arms: Active, 1
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
This study examined the benefit of continued treatment with an antidepressant medication, sertraline, in adolescents with depression who improved on sertraline acutely. We hypothesize that adolescents who remained on sertraline long term were less likely to have a recurrence of depression compared to those on placebo.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial of maintenance treatment of sertraline in adolescents aged 13-19 with depression.

Subjects Subjects aged 13-19 were recruited, over 18 months, at mood disorders clinics in 3 tertiary care centres across Canada. Informed consent was obtained from eligible and interested subjects and parents (if subject <16 years of age). Subjects were eligible for entry into the study if they had a diagnosis of Major Depression determined from both clinical interview and the Schedule for Affective Disorders and Schizophrenia for Children (K-SAD-PL) and scored > 16 on the first 17 items of the 29-item Hamilton Rating Scale for Depression (HAM-D). Subjects were excluded if they had past or current hypomanic or manic episode, current psychotic symptoms, substance dependence in the last 3 months, significant medical condition that would contra-indicate the use of antidepressants or that if untreated may require medical attention, pregnancy, or past treatment with sertraline for major depression.

Interventions and Procedures There were 3 phase to the study: 1) a 12-week acute phase, 2) a 24-week continuation phase, and 3) a 52-week maintenance phase. In general, subjects were assessed every 2 weeks throughout the study except during the first 4 weeks of the maintenance phase when they were seen or contacted weekly. In the continuation and maintenance phases, every 2nd visit was conducted in person while the other assessments could be conducted either by telephone or in person.

Initial sertraline dose during the acute phase was either 25 mg or 50 mg daily with increases of 25 to 50 mg every 2 weeks at the treating clinicians' discretion, up to a maximum of 200 mg daily. For responders who entered the continuation phase and had some re-emergence of symptoms without relapse, dose increases with sertraline were permitted every 2 weeks to a maximum dose of 200 mg daily but only during the first 8 weeks of the continuation phase. If a subject experienced side effects, one dose decrease was permitted in the first 8 weeks of the continuation phase. Subjects who maintained response during continuation were then randomized to continue sertraline or to take placebo. In the placebo group, sertraline was tapered by 25% of the initial dose every week for the first 4 weeks of the maintenance phase. During the maintenance phase, no treatment changes were permitted.

Subjects who responded to acute phase treatment, defined as 2 consecutive HAMD < 9 and greater than a 50% reduction in HAM-D score within 12 weeks, were offered entry into the continuation phase. Inter-rater reliability for the HAM-D was tested annually with site project coordinators and research assistants. Further training and evaluation were implemented until the inter-rater reliability was 0.8 or greater. Relapse during the continuation and recurrence during maintenance phases were determined according to the clinical judgement of the treating physician that the major depression had recurred or an intervention beyond what was permitted by the study protocol was required.

Adverse events were collected using the Common Adverse and Side Effects Scale. The scale was administered every 2 weeks during the acute phase and every 4 weeks during the continuation and maintenance phase.

Blinding and Randomization Randomization was conducted by the study pharmacist using a computer generated randomization schedule. Subjects, clinicians and research staff remained blinded to treatment during the randomization phase. All statistical analyses were conducted by an independent statistician blinded to patient allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-19
* Diagnosis of Major Depression

Exclusion Criteria:

* History of mania/hypomania
* Current psychotic symptoms
* Substance dependence
* Medical conditions (contraindication for sertraline)
* Pregnancy
* Past treatment with sertraline

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 1997-07

PRIMARY OUTCOMES:
recurrence of depression | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Levitt, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - UBC, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia

REFERENCES:
- [Derived] Cheung A, Kusumakar V, Kutcher S, Dubo E, Garland J, Weiss M, Kiss A, Levitt A. Maintenance study for adolescent depression. J Child Adolesc Psychopharmacol. 2008 Aug;18(4):389-94. doi: 10.1089/cap.2008.0001. PMID 18759650